CLINICAL TRIAL: NCT04430803
Title: The Effects of Six-month Hydrogen-rich Water Intake on Molecular and Phenotypic Biomarkers of Aging in Men and Women Aged 70 Years and Over: a Randomized-controlled Trial
Brief Title: Hydrogen-rich Water for Molecular and Phenotypic Biomarkers of Aging
Acronym: H2AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 281048E-HRW/2020
Record Dates: First submitted 2020-06-07; First posted 2020-06-12 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen-rich water (Experimental): Hydrogen-rich water (Rejuvenation, HRW Natural Health Products Inc.)
  * 8 ppm of hydrogen
  * Administered one dose two times per day on an empty stomach in the morning and at the evening
  Interventions: Dietary Supplement: Hydrogen-rich water
- Control water (Placebo Comparator): Tap water
  * 0 ppm of hydrogen
  * Administered one dose two times per day on an empty stomach in the morning and at the evening
  Interventions: Other: Control Water

INTERVENTIONS:
Dietary Supplement: Hydrogen-rich water — A tablet that produces hydrogen dissolved in a glass of water
  Arms: Hydrogen-rich water
Other: Control Water — A glass of tap water
  Arms: Control water

SUMMARY:
This study evaluates the effects of six-month hydrogen-rich water intake on molecular and phenotypic biomarkers of aging in men and women aged 70 years and over.

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years
* Free of acute disorders

Exclusion Criteria:

* History of dietary supplement use during the past 4 weeks

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in TeloTAGGG Telomerase PCR activity in serum | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months

SECONDARY OUTCOMES:
Change in DNA methylation | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in blood concentration of advanced glycation end product | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in lipid peroxidation | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in serum FGF21 | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in serum TET2 | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in ADAS-Cog score (0-70 scale, higher scores indicating greater cognitive impairment) | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in facial wrinkling (0-100 scale; higher scores mean worse outcome) | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in maximal oxygen uptake estimated by step-in-place test | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- FSPE Applied Bioenergetics Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xia X, Chen W, McDermott J, Han JJ. Molecular and phenotypic biomarkers of aging. F1000Res. 2017 Jun 9;6:860. doi: 10.12688/f1000research.10692.1. eCollection 2017. PMID 28663789
- [Derived] Zanini D, Todorovic N, Korovljev D, Stajer V, Ostojic J, Purac J, Kojic D, Vukasinovic E, Djordjievski S, Sopic M, Guzonjic A, Ninic A, Erceg S, Ostojic SM. The effects of 6-month hydrogen-rich water intake on molecular and phenotypic biomarkers of aging in older adults aged 70 years and over: A randomized controlled pilot trial. Exp Gerontol. 2021 Nov;155:111574. doi: 10.1016/j.exger.2021.111574. Epub 2021 Oct 1. PMID 34601077